CLINICAL TRIAL: NCT05644652
Title: Effect of Nordic Walking on Gait-asymmetry Patterns in Children With Hemiparesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amira Mahmoud Abd-elmonem, Assist Prof. Physiacl therapy for pediatric department, faculty of physical therapy , Cairo university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Nordic walking
Record Dates: First submitted 2022-09-29; First posted 2022-12-09 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Cerebral Palsy
Keywords: Cerebral palsy; gait; spatio-temporal gait parameters; unilateral cerebral palcy; Nordic walking
MeSH Terms: conditions — Cerebral Palsy | interventions — Nordic Walking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Experimental): 15 Children in this group will receive a designed physical therapy program for 60 minutes per session, three times a week, for three consecutive months.
  Interventions: Other: designed physical therapy program
- Nordic walking group (Experimental): Children in this group will receive the same designed physical therapy program for 60 minutes per session, three times a week, for three consecutive months. while the Nordic walking training for 20 minutes will replace the functional gait training.
  Interventions: Other: designed physical therapy program; Other: Nordic walking

INTERVENTIONS:
Other: designed physical therapy program — it will be applied for for 60 min weekly for 3 successive months in the form of three sets of exercises (15minutes each) as follows:
  * Flexibility exercises to restore joint mobility of soft tissues.
  * Static and dynamic balance exercises
  * Functional strengthening exercises.
  * Functional gait training.
Other: Nordic walking — it will be conducted according to the guidelines of the International Nordic Walking Federation
  Arms: Nordic walking group

SUMMARY:
Nordic walking is a physical activity consisting of walking with poles similar to ski poles. The poles are designed for the purpose of activating the upper body during walking. The poles are equipped with rubber or spike tips and the walking itself resembles.

DETAILED DESCRIPTION:
Compared to normal walking in Nordic walking there is a stronger involvement of the upper body. Furthermore, by using the poles, the muscles in the upper body can be activated, and the length of each step taken is supposedly increased, resulting in a faster gait .

ELIGIBILITY:
Inclusion Criteria:

* Their age will range from 6-10 years, from both sexes.
* Level I, II and III of gross motor functional classification system (GMFCS) (Jooyeon et al., 2011)
* Grade 1 and 1+ spasticity according to the Modified Ashworth Scale (MAS). (Cloptonetal et al., 2005).

Exclusion Criteria:

* Uncontrolled epilepsy.
* Mental retardation or autistic features.
* Significant visual or auditory problems according to medical reports (audio-vestibular and ophthalmic examination),
* Structural or fixed soft tissue deformities of the lower and/or upper extremities.
* Neurological or orthopedic surgery in the past 12 months in the lower and/or upper extremities.
* Botox injection in the lower and/or upper extremities in the past 6 months.

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Assessment of gait | after 3 successive months
  The gait parameters will be assessed by kinovea software. Kinovea, free 2D motion analysis software, was created in 2009 via the non-profit collaboration of several researchers, athletes, coaches and programmers from all over the world. It enables the analysis of distances, angles, coordinates and spatial-temporal parameters frame by frame from a video recording. These measurements can be made from different perspectives, since the software carries out calibrations in non-perpendicular planes to the camera-object line analyzed. spatio-temporal parameters will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Emam H El-negamy, Phd, Study Chair — Cairo university, faculty of physical therapy; Maricha A Nashed, B.Sc., Principal Investigator — Cairo university, faculty of physical therapy
Locations (1):
- Cairo University, Giza, Egypt

REFERENCES:
- [Derived] Nashed MA, Elnegmy EH, El-Tohamy AM, Abd-Elmonem AM. Efficacy of Nordic Walking Versus Conventional Gait Training on Gait Asymmetry Patterns in Children With Hemiparesis. Physiother Res Int. 2026 Jan;31(1):e70139. doi: 10.1002/pri.70139. PMID 41346090